CLINICAL TRIAL: NCT04493697
Title: Using Time Varying Non-Invasive Neuromodulation to Improve Neurovascular Status in Parkinson's Disease
Brief Title: Using Neuromodulation to Improve Parkinson's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Device provider has requested withdrawal citing modifications needed for study integrity.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00067408WD
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Motor/Non-Motor Symptoms; Neurovascular Symptoms
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: All participants will receive a ThermoNeuroModulation device for in-home use. Participants will be randomized to either the active or placebo treatment arm.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The device uses a bar code reader to import a prescription waveform. The use of the bar code aids blinding during randomization since the QR code is not readable by study members.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental 1 (Active Comparator): A ThermoNeuroModulation device will be worn by the participant that delivers warm waveforms in one ear (42 °C) and cool waveforms (17 °C) in the other ear.
  Interventions: Device: Experimental 1
- Experimental 2 (Placebo Comparator): A ThermoNeuroModulation device will be worn by the participant that will neither warm nor cool.
  Interventions: Device: Experimental 2

INTERVENTIONS:
Device: Experimental 1 — A ThermoNeuroModulation device will be worn by the participant that delivers warm waveforms in one ear (42 °C) and cool waveforms (17 °C) in the other ear.
  Arms: Experimental 1
Device: Experimental 2 — A ThermoNeuroModulation device will be worn by the participant that will neither warm nor cool.
  Arms: Experimental 2

SUMMARY:
This study is a single-site, double-blinded, placebo-controlled, randomized clinical trial designed to elucidate mechanism(s) of action for symptomatic benefits observed in Parkinson's disease (PD) patients treating twice daily time-varying caloric vestibular stimulation treatment using a solid-state device. Study participants will self-administer treatments in the home setting over a period of 12 weeks. Changes in cerebral blood flow perfusion, cerebrovascular reactivity and functional connectivity between the pre-treatment baseline and the end of the treatment period will be monitored and will be compared to changes in validated standardized clinical measures of motor and non-motor symptoms in PD. The durability of effects will be evaluated at a post-treatment assessment conducted five weeks after treatment cessation.

DETAILED DESCRIPTION:
A double-blinded, placebo-controlled randomized trial will explore the effects of time-varying caloric vestibular stimulation (tvCVS) treatments on changes in biomarkers of neurovascular status (i.e. cerebral blood flow perfusion and cerebrovascular reactivity) as well as their relationship to clinical endpoints. Participants will be randomly allocated in a 1:1 ratio using block randomization by the clinical site. Participants will be trained in the clinic to self-administer device treatment and then will continue to self-administer the ~19-minute treatments twice daily for 12 weeks in the home. Individual stimulation sessions will be spaced a minimum of 1 hour apart. Outcome measures will be administered at the baseline, the end of the 12-week treatment period and at 5 weeks post-treatment. Study participants will continue to take their approved Parkinson's disease (PD) medications throughout the study and will maintain patterns of usage throughout.

Previous evidence for efficacy demonstrated therapeutic gains as an adjuvant for standard of care treatment. Consistent with these observations, all outcome measures will be evaluated when study participants are in the on-medication state and at the same time relative to the last dose of anti-Parkinsonian medication across all assessments. Clinical measures will be captured at the baseline, at the end of treatment period, and again five weeks after cessation of treatment. Most of the planned clinical measures including the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) parts I, II, and IV, the Non-Motor Symptom Scale for PD (NMSS), the Montreal Cognitive Assessment (MoCA), the Parkinson's Anxiety Scale, the Geriatric Depression Scale, the Epworth Sleepiness Scale, and the Functional Assessment of Chronic Illness Therapy- Fatigue are suitable for virtual collection. Case report forms (CRFs) for the patient reported outcomes will be provided to study participants via standard mail. At the end of each virtual visit, participants will be asked to complete these forms and bring them to the clinic the next day when they come for their in-clinic visit. In the case where an in-clinic visit may not be possible, participants will be asked to show completed forms to the coordinator via the telemedicine platform to confirm completeness, and forms will be collected at the next in-person visit or can be mailed in by the participant.

The full MDS- UPDRS part III and the Timed Up and Go will be administered in the clinic. However, a modified MDS-UPDRS part III (excluding items related to rigidity or postural instability) will also be administered through the telemedicine platform. This measure will serve as backup for cases where participants may be unable to come into the clinic for regularly scheduled assessment (e.g. due to COVID-19 containment measures).

ELIGIBILITY:
Inclusion Criteria:

* Must be 21-85 years old.
* Diagnosed with Parkinson's Disease (meeting UK PD Society Brain Bank criteria)
* Responsive to oral DRT (dopamine replacement therapy) for a minimum of 3 years and on a stable dose of therapy
* Must be able to voluntarily give written informed consent
* Must have ability to reliably use the investigational device
* Must be able to understand and complete all assessments (provided in English only) within a given on-state period
* Must be willing and able to undertake a ~1 hour imaging session in a MRI magnet with a head coil in place during 3 separate clinic visits.
* Must have a home partner and/or regular caregiver
* Must have capability to complete assessments using telemedicine platforms.
* Must demonstrate moderate burden of motor symptoms and non-motor symptoms in PD ( MDS-UPDRS part II >12 and MDS-UPDRS part I scores >10)

Exclusion Criteria:

* Pregnant women.
* Have experienced a heart attack, angina or stroke within the past 12 months,
* Use of medications that regulate heart rate
* Have a history or prior diagnosis of dementia or adjusted score ≤ 20 on the Montreal Cognitive Exam at the baseline visit.
* Those receiving deep brain stimulation
* Treated with a pump for continuous delivery of DRT (Dopamine replacement therapy)
* Use of Apomorphine rescue
* Works night shifts
* Have a major concomitant illness or illnesses including cancer or disease of the cardiovascular, respiratory and/or renal systems
* Has history or evidence of unstable mood disorder, or responds affirmatively to question #9 on the BDI-II (any score > 0 on suicidal thoughts or wishes). Participants that respond affirmatively to this question should receive a referral for mental health counseling according to the mandates of the IRB or ethics review committee.
* Those with hearing aids or cochlear implants, chronic tinnitus, temporomandibular joint disease
* Those who have persistent negative sequela of a traumatic brain injury
* Those who have been diagnosed with another neurological illness with the exceptions of restless leg syndrome and REM behavioral sleep disorder
* Those with a recent history of substance abuse and/or dependence (alcohol or other drugs)
* Those who have a diagnosed vestibular dysfunction and/or balance dysfunction
* Those who have had eye surgery within the previous three months or ear surgery within the previous six months
* Those who have inner ear pathology, such as active and/or frequent ear infections or reported damage to the tympanic membrane or have labyrinthitis
* Those who have contraindications for MRI imaging, such as metal implants or a pacemaker that would preclude the MRI scan
* Those who have participated in another clinical trial within the last 30 days or are currently enrolled in another clinical trial
* Those who are taking antiemetics chronically (more than 2 times per week, consistently) due to known interference with the vestibular response to caloric stimulation

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Neuroimaging | Baseline
  Brain data will be acquired with Siemens MAGNETOM Skyra 3T MRI - range measured by statistically significant change in cerebral blood flow (CBF) measured in units of mL/100g/min
Neuroimaging | Week 12
  Brain data will be acquired with Siemens MAGNETOM Skyra 3T MRI - range measured by statistically significant change in cerebral blood flow (CBF) measured in units of mL/100g/min
Neuroimaging | Week 17
  Brain data will be acquired with Siemens MAGNETOM Skyra 3T MRI - range measured by statistically significant change in cerebral blood flow (CBF) measured in units of mL/100g/min
Transcranial Doppler Sonography | Baseline
  Non-invasive ultrasound used to examine blood circulation within the brain - range measured by statistically significant change in mean cerebral blood flow velocity (cm/s)
Transcranial Doppler Sonography | Week 12
  Non-invasive ultrasound used to examine blood circulation within the brain - range measured by statistically significant change in mean cerebral blood flow velocity (cm/s)

SECONDARY OUTCOMES:
MDS-Unified Parkinson's Disease Rating Scale | Baseline, Week 12, Week 17
  Used to follow the longitudinal course of symptoms of Parkinson's disease - Each parkinsonian sign or symptom is rated on a 5-point Likert-type scale (ranging from 0 to 4), with higher scores indicating more severe impairment. The maximum total UPDRS score is 199, indicating the worst possible disability from PD
Timed Up and Go Test | Baseline, Week 12, Week 17
  To determine fall risk and measure the progress of balance, sit to stand and walking (ranging from ≤10 seconds as normal to 30 seconds as high fall risk).
Montreal Cognitive Assessment | Baseline, Week 12, Week 17
  Cognitive screening test - range from zero to 30, with a score of 26 and higher generally considered normal.
Non-Motor Symptom Scale | Baseline, Week 12, Week 17
  Scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease - 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The NMSS measures the severity and frequency of non-motor symptoms across nine dimensions - the total NMSQuest score significantly increased with disease severity and duration meaning that the number of individual non-motor symptoms reported by our patients increases as the disease progresses.
Geriatric Depression Scale | Baseline, Week 12, Week 17
  A self-report measure of depression in older adults - Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Parkinson's Anxiety Scale | Baseline, Week 12, Week 17
  Anxiety assessment - The PAS is a 12-item observer or patient-rated scale with three subscales, for persistent, episodic anxiety and avoidance behavior - There is a maximum total score of 48. Higher scores indicate great experiences of anxiety.
Epworth Sleepiness Scale | Baseline, Week 12, Week 17
  A self-administered questionnaire to assess the daytime sleepiness - The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Functional Assessment of Chronic Illness Therapy - Fatigue - | Baseline, Week 12, Week 17
  A tool to help manage chronic illness - The responses to the 13 items on the FACIT fatigue questionnaire are each measured on a 4-point Likert scale. Thus, the total score ranges from 0 to 52. High scores represent less fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Christopher T Whitlow, MD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No